CLINICAL TRIAL: NCT01490593
Title: Canadian Eye Injury Registry
Acronym: CEIR
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian National Institute for the Blind (Other)
Responsible Party: Sponsor
Other Study IDs: R-11-079; 17853e (Other: REB)
Record Dates: First submitted 2011-06-29; First posted 2011-12-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Eye Injuries
Keywords: Canadian; Eye; Injury; Registry
MeSH Terms: conditions — Eye Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Eye Injuries: The database is being established to record the number and types of eye injuries occurring in Canada. Thus there is only one cohort group, individuals who have sustained an eye injury.
  Interventions: Behavioral: Public Health strategies

INTERVENTIONS:
Behavioral: Public Health strategies — It is hoped that by recording of the data (i.e. locations and mechanisms of eye injuries), we may be able to develop public health strategies to prevent further injuries. For example, encouraging more visor wear in hockey games if we notice increased prevalence of hockey eye injuries with no visor.
  Other Names: CEIR

SUMMARY:
The purpose of this study is to establish an eye injury registry to assess the mechanisms and outcomes of significant eye injuries occurring in Canada. The epidemiologic data will determine where public health strategies should be directed to prevent future eye injuries.

DETAILED DESCRIPTION:
Currently there is no established database or recording system of eye injuries occurring in Canada. Estimates place the figure at approximately 100000 significant eye injuries occurring in our country every year. This represents a large public health and long-term disability challenge. Lost productivity of working-age individuals with vision loss amounts to $4.4 billion annually in Canada, part of which is due to eye injury. By recording the types, locations, and outcomes of significant eye injuries, it is hoped improved public health strategies may be established to prevent further ones. The need for such a database has been recognized by the Ivey Eye Institute, the Canadian National Institute for the Blind (CNIB) and the Canadian Ophthalmological Society (COS).

The United States Eye Injury Registry (USEIR) has been in existence for greater than 20 years. Through their database they have recorded thousands of eye injuries which has led to public health interventions through their various ocular societies. They have also established a standardized reporting system and ocular trauma score which has improved diagnosis and prognosis of eye injuries. This system has been used in many countries as a standardized reporting scheme for eye injuries.

It is hoped that through a pilot recording system established in London a framework for a national reporting system will develop. The objective is to use the standardized reporting system of the USEIR to report Canadian eye injuries.

The time frame for outcome measures will be 6 months. The patients will be followed along for this amount of time to assess there visual outcomes. No further follow up after 6 months will be undertaken for the purpose of the registry.

The hypothesis is that by recording the type and outcome of eye injuries, a better understanding of mechanisms and location of these injuries in Canada will occur. Subsequent public health interventions can then be made in conjunction with the CNIB and COS to improve eye health in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who experiences an acute eye injury that has or has the potential to compromise the integrity of the eye. These are serious eye injuries resulting in permanent and significant (i.e. measurable or observable on routine eye examination) structural or functional change to the eye. Separate reports are to be filed for each eye involved in bilateral injuries.

Exclusion Criteria:

* Based on the standard of the United States Eye Injury Registry
* Mild ocular contusions
* Subconjunctival hemorrhage
* Superficial abrasions by themselves usually would not meet the criterion of serious and/or reportable injuries.
* The exclusion of these injuries will depend on the clinical judgement of the reporting physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals who have sustained a serious eye injury in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Number and type of eye injuries occurring in Canada | 6 months
  To record and determine the types and epidemiologic data of eye injuries in Canada.

SECONDARY OUTCOMES:
Ocular Trauma Score | 6 months
  To determine the correlation between the ocular trauma score as defined by the American Society of Ocular Trauma and the actual visual outcomes of Canadian Eye Injury patients

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Hooper, MD, Principal Investigator — The University of Western Ontario - Ivey Eye Institute
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada

REFERENCES:
- [Background] Kuhn F, Morris R, Witherspoon CD, Mann L. Epidemiology of blinding trauma in the United States Eye Injury Registry. Ophthalmic Epidemiol. 2006 Jun;13(3):209-16. doi: 10.1080/09286580600665886. PMID 16854775